CLINICAL TRIAL: NCT02496832
Title: An Exploratory Study of Hypoxia Imaging Using 18F-FAZA-PET in Advanced Pancreatic Cancer Patients Being Treated With Gemcitabine + TH-302/Placebo (MAESTRO: EMR200592-001)
Brief Title: A Study of Hypoxia Imaging in Advanced Pancreatic Cancer Patients Being Treated With Gemcitabine and TH-302 or TH-302 Placebo
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never initiated
Sponsor: University Health Network, Toronto (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Faza-Maestro
Record Dates: First submitted 2014-05-28; First posted 2015-07-14 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Pancreatic Adenocarcinoma; Advanced Disease; Metastatic Disease
Keywords: Hypoxia; 18F-FAZA; 18F-Fluoroazomycin arabinoside; Positron emission tomography; PET; Participating in study EMR200592-001
MeSH Terms: conditions — Neoplasm Metastasis; Hypoxia | interventions — fluoroazomycin arabinoside

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FAZA PET-CT scan (Experimental): FAZA PET-CT imaging within 14 days of treatment from the EMR200592-001 study.
  FAZA PET-CT imaging about 5 weeks after start of treatment from the EMR200592-001 study.
  Interventions: Drug: 18F-Fluoroazomycin arabinoside

INTERVENTIONS:
Drug: 18F-Fluoroazomycin arabinoside
  Other Names: 18F-FAZA; [18F] FAZA

SUMMARY:
Researchers are looking for better ways of diagnosing and treating pancreatic cancer. It is believed that looking for low levels of oxygen (hypoxia) in tumours may give a better understanding of how certain tumours grow or respond to certain treatments. This study will look at hypoxia in pancreatic tumours while participants are receiving treatment with the combination of gemcitabine and TH-302/placebo in the EMR 200592-001 clinical research study.

This study will use positron emission tomography (PET) scans to look at hypoxia in tumours. PET is an imaging test that can be used to measure hypoxia in tumours. For this study, a radioactive tracer called Fluoroazomycin Arabinoside (FAZA) will be used to "label" areas of hypoxia in tumours. Determining the levels of hypoxia in tumour tissue using FAZA-PET scans and comparing these levels with the patient's response to treatment with gemcitabine and TH-302/placebo for pancreatic cancer may help the researchers to determine the relationship between hypoxia and response to this treatment.

The main purpose of this study is to see how useful looking at hypoxia in tumours are when they are done at different centres.

ELIGIBILITY:
Inclusion Criteria:

* Have consented to participating on the first-line Gemcitabine + TH-302/placebo (study number EMR200592-001) study
* Age 18 years or older
* Cytologic/histologic diagnosis of pancreatic adenocarcinoma
* Advanced stage pancreatic cancer: locally advanced or metastatic.
* No prior chemotherapy for advanced/metastatic disease. Adjuvant chemotherapy allowed if completed > 6mths from study entry. Prior radio-sensitizing doses of 5-FU or gemcitabine also allowed.
* ECOG performance status 1 or less
* Adequate end organ and marrow function
* Measureable or non-measureable disease by RECIST 1.1
* Female patients of child-bearing potential must have a negative serum pregnancy test (BhCG) and must agree to abstinence or use adequate contraception for the duration of the study
* Disease-free period of more than 5 years from prior malignancies other than pancreas (except curatively treated basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix and ductal carcinoma in situ (DCIS) breast disease).
* Ability to provide written informed consent
* Must be able to lie flat comfortably for 30 to 60 min to complete imaging study

Exclusion Criteria:

* Inability to lie supine for 30 to 60 minutes
* Concurrent second primary
* Life expectancy of less than 12 weeks
* On treatment with disulfiram (antabuse) due to [18F]FAZA injection containing up to 10% (v/v) ethanol in PBS (phosphate-buffered saline)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Expected number of similar quality scans produced compared to actual number of similar quality scans produced using the same method is less than 15%. | 2 years
Number of enrolled patients that complete all required scans compared to total number of patients enrolled in the study is at least 70%. | 2 years
Range of tumor hypoxia in patients with pancreatic cancer that had not received prior treatment. | 2 years

SECONDARY OUTCOMES:
Compare the changes in tumor hypoxia before chemotherapy treatments and after chemotherapy treatments. | 2 years
Compare the changes in tumor hypoxia with response to chemotherapy treatments. | 2 years
Evaluate how FAZA is taken in by different tumor types within individual patients. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Neesha Dhani, M.D., Principal Investigator — Princess Margaret Cancer Centre